CLINICAL TRIAL: NCT07090798
Title: Applied Virtual Reality Techniques In Musculoskeletal Assessment Of Cervical Ergonomic Disorders Among Dentists
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Feyza Sule BADILLI HANTAL, asst.prof, Yeditepe University
Other Study IDs: Virtual
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cervical Pain
Keywords: dentists, cervical pain, virtual reality, clinical, physical, postural, functional, assessment
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Static Head posture — After the participant sit down and put on the VR glasses, the VR will detect how many degrees the head position has displaced from the neutral position (X= 0, Y = 0, Z = 0). The x, y and z describe the head alignment, and in the table (3.3), they explain the 3D axis (X, Y, Z). Also in fig 3.3 the participant's head is in X=5.027058 Y=2.466827 Z=2.93206, which explains the degree of deviation from the neutral position.
Diagnostic Test: Angular distance "ROM" — Cervical range of motion assessment is achieved through virtual reality. After detecting the static head posture, Participants will be asked to flex their necks as far as possible toward their chins and anterior chests. Then elevate the head to the neutral and extend the neck to the most tolerable range. Following that, he/she performs maximal neck side-bending in both directions along the coronal plane. Lastly, each participant is required to return the neck to an upright position for the examination of the maximum angle of neck rotation by "turning the chin toward the right and then left shoulders" without shrugging the shoulders. All of the tests will be repeated three times, and the averaged values of neck movement in each direction will be taken for analysis

SUMMARY:
This study aims to evaluate the effectiveness of a virtual reality (VR)-based assessment system in identifying clinical, physical, and functional impairments related to neck pain and musculoskeletal disorders (NPMSDs) among dentists. Forty dentists with neck pain were assessed using a structured protocol including sociodemographic data collection, the Neck Disability Index, VR-based measurements of head posture and cervical motion (with and without pain), and muscle strength testing via a digital dynamometer. The study investigates the predictive value of VR-derived parameters-such as head alignment, range of motion, and movement time and degree-with regard to pain and functional status. Findings suggest that virtual reality can serve as an objective, non-invasive tool for evaluating cervical spine health in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age group from 29 to 60 years.
2. All the participants with neck pain, with or without referral to the upper limb, longer than 4 weeks.
3. Etiology of mechanical neck pain due to dentists work.

Exclusion Criteria:

* 1. Suffering from visual or vestibular disorders. 2. chronic intake of drugs which may alter pain or performance . 3. after whiplash injury .

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Licensed dentists currently working in clinical settings who report neck pain related to musculoskeletal disorders. All participants were recruited from the Faculty of Health Sciences at Yeditepe University. The sample includes both male and female dentists aged between 25 and 40 years, with a minimum of one year of clinical work experience. Participants were experiencing varying levels of neck pain and disability but were otherwise healthy and capable of completing the assessment procedures.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Neck Disability index | Baseline (single time)
  The Neck Disability Index is a ten-item self-reported questionnaire describing daily life, pain, and concentration. Each item is rated on a score from 0-5, with 0 indicating no disability and 5 indicating extreme disability. To be clinically meaningful, there must be a minimum clinically important difference (MCID) of 5 points, at least, from a total of 50 (Table 3.2). Many studies have confirmed that the NDI has a high degree of validity and reliability. The NDI has also been used as an outcome measure in a number of studies involving the treatment of neck pain and patients with whiplash injury

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sterling M, Hendrikz J, Kenardy J. Compensation claim lodgement and health outcome developmental trajectories following whiplash injury: A prospective study. Pain. 2010 Jul;150(1):22-28. doi: 10.1016/j.pain.2010.02.013. Epub 2010 Mar 21. PMID 20307934
- [Result] Cunha AC, Burke TN, Franca FJ, Marques AP. Effect of global posture reeducation and of static stretching on pain, range of motion, and quality of life in women with chronic neck pain: a randomized clinical trial. Clinics (Sao Paulo). 2008 Dec;63(6):763-70. doi: 10.1590/s1807-59322008000600010. PMID 19060998